CLINICAL TRIAL: NCT00694759
Title: Cortisol Regulation in Polycystic Ovary Syndrome
Brief Title: Cortisol Regulation in Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Bethany Klopfenstein, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OHSUIRB00002532
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; insulin; PCOS; cortisol regulation; regulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Pioglitazone will be given to women with PCOS. After one month and six months of therapy, measure (a) 24-hour CPR, ACTH, free cortisol, and CBG, (b) adipocyte, liver, and whole body HSD 1 activity, and (c) insulin sensitivity, visceral fat, and androgen levels.
  Interventions: Drug: pioglitazone
- B (Active Comparator): Metformin will be given to women with PCOS. After one month and six months of therapy, measure (a) 24-hour CPR, ACTH, free cortisol, and CBG, (b) adipocyte, liver, and whole body HSD 1 activity, and (c) insulin sensitivity, visceral fat, and androgen levels.
  Interventions: Drug: metformin
- C (Placebo Comparator): Placebo will be given to women with PCOS. After one month and six months of therapy, measure (a) 24-hour CPR, ACTH, free cortisol, and CBG, (b) adipocyte, liver, and whole body HSD 1 activity, and (c) insulin sensitivity, visceral fat, and androgen levels.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pioglitazone — 30 mg for 2 weeks, then 45 mg daily
  Other Names: Actos
  Arms: A
Drug: metformin — 500mg twice daily for 1 week, then 1000 mg twice daily
  Other Names: Glucophage; Glucophage XR
  Arms: B
Drug: placebo — capsule twice daily
  Arms: C

SUMMARY:
The purpose of this study is to determine if insulin resistance (how well the body uses insulin and clears sugar) can affect cortisol levels in normal healthy women and women with polycystic ovary syndrome of all body weights.

DETAILED DESCRIPTION:
PCOS is a common clinical problem affecting young women, characterized by oligomenorrhea and hyperandrogenism. Central obesity and insulin resistance are also prominent features of PCOS, and in addition are important risk factors for development of hypertension, hyperlipidemia and atherosclerotic heart disease. Previous studies have suggested that cortisol is dysregulated in PCOS, primarily through increased hypothalamic-pituitary-adrenal (HPA) axis activity and enhanced cortisol secretion. Increased adrenocorticotropic hormone (ACTH) secretion could also potentially lead to elevated adrenal androgen production in PCOS. Techniques used in previous studies have been inconsistent, however, and a link between increased HPA axis activity and the phenotypic changes in PCOS has not been clearly demonstrated. Cortisol is also produced from cortisone in peripheral adipose tissue by the enzyme 11beta-hydroxysteroid dehydrogenase type 1 (HSD 1), suggesting another potential point of dysregulation that may contribute to central obesity and insulin resistance in PCOS. Further investigation of both central and peripheral regulation of cortisol is necessary to better understand the pathophysiology of PCOS.

Specific Aim 1: To perform a cross-sectional study of women with PCOS and normal controls matched for age and body mass index, and measure insulin sensitivity and visceral fat, as well as (a) 24-hour CPR, ACTH, free cortisol, and cortisol binding globulin (CBG), (b) adipocyte, liver, and whole body HSD 1 activity, and (c) androgen levels.

Specific Aim 2: To prospectively administer pioglitazone or metformin to women with PCOS in a placebo-controlled trial, and after one month and six months of therapy measure (a) 24-hour CPR, ACTH, free cortisol, and CBG, (b) adipocyte, liver, and whole body HSD 1 activity, and (c) insulin sensitivity, visceral fat, and androgen levels.

ELIGIBILITY:
Inclusion Criteria (Healthy controls):

* Healthy
* At lifetime maximal weight
* Weight stable for at least 6 months prior to study entry
* Willing to commit to not making significant changes to their diet or daily activities while enrolled.
* Premenopausal
* Have regular menstrual cycles
* No evidence of hirsutism

Additional Inclusion Criteria (Subjects with PCOS):

* Clinical findings of amenorrhea or oligomenorrhea dating from menarche
* Clinical and/or biochemical evidence of hyperandrogenism
* Exclusion of related disorders

Exclusion Criteria (Healthy controls):

* Less than 18 years of age
* Exercise > 30 minutes/day, 3 times a week
* Smokers
* Heavy alcohol drinkers (> 2 drinks/day)
* Type 2 diabetes
* Medical diagnoses including heart disease and cancer
* Psychiatric illness (i.e.depression, psychosis, bipolar, schizophrenia)
* Body weight > 136 kg
* Pregnant
* Endocrine diseases affecting body composition or androgen levels

Additional Exclusion Criteria (Subjects with PCOS):

* Laboratory evidence of hyperprolactinemia, thyroid dysfunction, or 21-hydroxylase-deficient nonclassic CAH
* Contraindication to pioglitazone (i.e. CHF, impaired liver function, anemia, depressed leukocyte counts, pulmonary disease, known sensitivity to thiazolidinediones.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The comparison of body surface area adjusted cortisol production rate (CPR/BSA) before insulin sensitizing therapy in women with PCOS. | Before 6 months of insulin sensitizing therapy
The comparison of body surface area adjusted cortisol production rate (CPR/BSA) after insulin sensitizing therapy in women with PCOS. | After 6 months of insulin sensitizing therapy

SECONDARY OUTCOMES:
Comparisons of 24-hour values for adrenocorticotropic hormone , free-cortisol, and cortisol binding globulin. | Before 6 months of insulin sensitizing therapy
Comparisons of 24-hour values for adrenocorticotropic hormone , free-cortisol, and cortisol binding globulin. | After 6 months of insulin sensitizing therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bethany J. Klopfenstein, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States